CLINICAL TRIAL: NCT04638621
Title: Precision Medicine for Dilated Cardiomyopathy-Cardiac Magnetic Resonance to Identify Early Family Phenotypes
Brief Title: Dilated Cardiomyopathy-Cardiac Magnetic Resonance (DCM-CMR) Ancillary Study
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ray Hershberger, Professor of Medicine, Human Genetics, and Cardiovascular Medicine, Ohio State University
Other Study IDs: 831408; R01HL148581-01A1 (NIH)
Record Dates: First submitted 2020-11-09; First posted 2020-11-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA, serum and plasma are collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Dilated Cardiomyopathy-Cardiac Magnetic Resonance (DCM-CMR) Study is an ancillary study from the parent study, DCM Precision Medicine Study. The rationale for the DCM-CMR study is to leverage cardiac magnetic resonance (CMR) imaging to detect earliest findings of DCM in the at-risk family members enrolled into the parent study.

DETAILED DESCRIPTION:
Dilated cardiomyopathy of unknown cause (DCM) is a major public health problem affecting more than a million people in the U.S. Most DCM is now known to have an underlying genetic basis. First-degree relatives (FDRs) of an individual with DCM are considered to be genetically at risk, particularly if they carry variants classified as pathogenic (P), likely pathogenic (LP) or uncertain significance (VUS) in DCM genes. Practice guidelines recommend that these FDRs undergo serial imaging because prompt intervention may avert advanced disease. While tissue damage is already well underway when DCM is manifest, myocardial tissue changes, termed "pre-DCM" herein, are known to precede adverse changes in myocardial structure and function. The investigators central hypothesis states that cardiac magnetic resonance (CMR) imaging may detect pre-DCM in individuals with increased genetic risk by identifying myocardial tissue changes prior to myocardial structural and functional changes. CMR measures of myocardial tissue characteristics, including late gadolinium enhancement and myocardial T1 mapping, have been histopathologically validated and have established diagnostic and prognostic value in DCM. Thus, the investigators specific hypotheses state that adverse CMR-based myocardial tissue characteristics will be associated with (1) A higher burden (number) of relevant variants (P, LP, VUS) in established DCM genes; and (2) Subsequent adverse changes in measures of cardiac structure and function. The investigators propose to leverage the DCM Precision Medicine Study, a multisite DCM Consortium study now with 1230 DCM patients (probands), balanced for race and sex, and their FDRs, most with no history of DCM. FDRs are cascade tested for relevant variants (P, LP, VUS) in DCM genes identified in probands. The investigators aim to (1) Estimate the associations between CMR-based myocardial tissue characteristics and the number (burden) of the proband's variants in DCM genes in at-risk FDRs. In 650 FDRs of probands with LP/P variants and/or VUSs, CMR scans will be completed at 9 participating DCM Consortium sites. The association between CMR-based myocardial tissue characteristics and the number of the proband's variants of each class (LP/P, VUS) carried by an at-risk FDR in a particular age group will be evaluated, adjusting for biologically relevant covariates. The investigators will also (2) Estimate the association between CMR-based myocardial tissue characteristics and subsequent changes in measures of cardiac structure and function in FDRs with normal baseline left-ventricular size and function. FDRs examined in Aim 1 will receive a second CMR exam 2.5 years after their baseline exam. The investigators will estimate the covariate-adjusted associations between baseline myocardial tissue characteristics and subsequent changes in CMR-derived measures of cardiac structure and function in groups defined by the most deleterious of the proband's variants carried (none, VUS, or LP/P). This study will validate a CMR-derived "pre-DCM" phenotype for FDRs who carry P or LP variants (established risk), and also provide preliminary evidence that some VUSs are biologically relevant.

ELIGIBILITY:
Inclusion Criteria:

1. The FDR's proband was enrolled in the DCM Precision Medicine Study at 1 of 9 participating sites, or exceptions granted by study PI.
2. The FDR's proband has had one or more variants identified, including P, LP and VUS.
3. The FDR is able report to one of the participating sites for study enrollment.
4. The FDR has no current contraindication for CMR (glomerular filtration rate (GFR) <30 mL/min/1.73 m2, non-compatible device implant, or allergy to gadolinium contrast).
5. The FDR has had no prior heart transplant.
6. The FDR is ≥18 years of age.
7. All races/ethnicity
8. Ability to give informed consent.
9. Ability to communicate in English.
10. Subject is not pregnant (CMR may be conducted 3-6 months post delivery)
11. Willingness to participate in a family-based study (subject willing to interact with OSU).

Exclusion Criteria:

1. Coronary artery disease (CAD) causing ischemic cardiomyopathy (> 50% narrowing, any major epicardial coronary artery).
2. Primary valvular disease.
3. Adriamycin or other cardiotoxic drug exposure.
4. Other forms of cardiomyopathy: Hypertrophic, Restrictive, or Arrhythmogenic Right Ventricular Dysplasia/Cardiomyopathy.
5. Congenital heart disease.
6. Other detectable causes of dilated cardiomyopathy, including sarcoid and hemochromatosis.
7. Other active multisystem disease, even if very rare, that may plausibly cause DCM (e.g., hypereosinophilic syndrome, cardiac involvement with connective tissue disease, Loeffler's endocarditis, endomyocardial fibrosis, etc) are excluded. Please call the PI to discuss if uncertain or not clear.
8. Severe and untreated or untreatable hypertension (systolic blood pressures routinely greater than 180 mm Hg and/or diastolic blood pressures greater than 120 mm Hg, and if resistant to multidrug treatment). This includes profound hypertension associated with other multisystem disease (e.g., scleroderma, other vasculitides, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 650 FDRs of probands from the parent study (DCM Precision Medicine Study) with no contraindication to CMR with contrast.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The association between CMR-derived tissue characteristics and the number (burden) of the proband's variants in DCM genes in at-risk first-degree relatives | The initial 2.5 years of the study.
  The burden of likely pathogenic or pathogenic variants in DCM genes in first-degree relatives and the association with worse values of CMR measures of myocardial tissue characterization will be analyzed, after controlling for biologically relevant covariates.
The changes in CMR tissue characterization over time in family members scanned for Outcome 1 who had normal left ventricular size and function | A subsequent 2.5 year time period
  The measures of myocardial tissue characterization in first-degree relatives will be evaluated in a follow up CMR exam, on average, at 2.5 years following a first DCM exam, to assess changes in myocardial structure and function, again analyzed in association with the burden of likely pathogenic or pathogenic variants in DCM genes.

CONTACTS AND LOCATIONS:
Overall Officials: Ray Hershberger, MD, Principal Investigator — Ohio State University; Karolina Zareba, MD, Principal Investigator — Ohio State University; Daniel Kinnamon, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States